CLINICAL TRIAL: NCT00020969
Title: Phase Two Multicenter Study Of Arsenic Trioxide In Patients With Myelodysplastic Syndromes
Brief Title: Arsenic Trioxide in Treating Patients With Myelodysplastic Syndromes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: CTI BioPharma (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CTI-1058; CDR0000068734 (Registry Identifier: PDQ (Physician Data Query)); UCLA-HSPC-010104701; NCI-G01-1971
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: refractory anemia; refractory anemia with ringed sideroblasts; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; atypical chronic myeloid leukemia, BCR-ABL1 negative; myelodysplastic/myeloproliferative neoplasm, unclassifiable
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders | interventions — Arsenic Trioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: arsenic trioxide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of arsenic trioxide in treating patients who have myelodysplastic syndromes.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the percentage of patients with low-risk myelodysplastic syndromes (MDS) who achieve a major hematologic improvement after treatment with arsenic trioxide.
* Determine the percentage of patients with high-risk MDS who achieve complete or partial remission or major hematological improvement after treatment with this drug.
* Determine the durability of responses in patients treated with this drug.
* Determine the duration of overall and progression-free survival of patients treated with this drug.
* Assess the quality of life of patients treated with this drug.
* Assess the toxicity profile of this drug in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to risk score (low risk vs high risk).

Patients receive arsenic trioxide IV 5 days a week on weeks 1-2. Treatment repeats every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients with stable disease or better may receive additional courses of treatment. Patients who achieve a complete remission (CR) should receive 2 additional courses of treatment after documentation of CR.

Quality of life is assessed at baseline, every 8 weeks during study, and then at 4 weeks after study completion.

Patients are followed at 4 weeks, every 3 months until completion of study treatment, and then annually thereafter.

PROJECTED ACCRUAL: A total of 30-110 patients (15-55 per stratum) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of myelodysplastic syndromes (MDS)

  * Refractory anemia (RA)
  * RA with ringed sideroblasts
  * RA with excess blasts (RAEB)
  * RAEB in transformation
  * Chronic myelomonocytic leukemia
* Low-risk MDS patients:

  * If serum erythropoietin less than 200 IU/mL, must have failed prior recombinant epoetin alfa (EPO) trial
* No prior acute myeloid leukemia

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* More than 3 months

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 2.5 times upper limit of normal (ULN)
* SGPT and SGOT no greater than 2.5 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* Absolute QT interval less than 460 msec in the presence of magnesium greater than 1.8 mg/dL and potassium greater than 4.0 mEq/L

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* At least 30 days since prior biologic therapy (except recombinant EPO in low-risk MDS patients)

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 30 days since prior radiotherapy

Surgery:

* Not specified

Other:

* At least 30 days since prior cytotoxic agents
* At least 30 days since prior investigational agents
* No prior arsenic trioxide

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-03 (Actual); Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott C. Stromatt, MD, Study Chair — CTI BioPharma
Locations (8):
- United States (8):
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Green Cancer Center at Scripps Clinic, La Jolla, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - St. Joseph Hospital Regional Cancer Center - Orange, Orange, California
  - Lynn Regional Cancer Center West, Boca Raton, Florida
  - Georgia Cancer Specialists - Northside Office, Atlanta, Georgia
  - Corpus Christi Cancer Center, Corpus Christi, Texas

REFERENCES:
- [Result] Schiller GJ, Slack J, Hainsworth JD, Mason J, Saleh M, Rizzieri D, Douer D, List AF. Phase II multicenter study of arsenic trioxide in patients with myelodysplastic syndromes. J Clin Oncol. 2006 Jun 1;24(16):2456-64. doi: 10.1200/JCO.2005.03.7903. Epub 2006 May 1. PMID 16651647